CLINICAL TRIAL: NCT04131205
Title: Role of Magnetic Resonance Imaging in Detection of Minimal Hepatic Encephalopathy
Brief Title: Role of MRI in Detection of Minimal Hepatic Encephalopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana, Faculty of Medicine (Other); Medical University of Graz (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Sebastian Stefanovic, MD, Clinical Investigator, University Medical Centre Ljubljana
Other Study IDs: HepaticEncephalopathy
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Liver Cirrhoses; Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Minimal Hepatic Encephalopathy: Patients with hyperammonemia and minimal hepatic encephalopathy
  Interventions: Diagnostic Test: Magnetic Resonance Imaging
- Control: Healthy controls
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — We will assess the role of magnetic resonance (MR) in mHE diagnosis with emphasis on multimodal imaging technique
  Other Names: Ammonia Levels; Child Pugh Score; West-Haven grade of Hepatic Encephalopathy

SUMMARY:
Introduction Liver cirrhosis (LC) is irreversible fibrosis of the liver (1) and it remains a public health problem. One of the complications of the cirrhosis is hepatic encephalopathy (HE) which is defined as brain dysfunction caused by liver insufficiency. Pathophysiological mechanisms of HE are complex and multifactorial. Recognition of beginning stages of HE, such as minimal HE (mHE) is of most importance.

Objectives and originality of the project Diagnosis of mHE can be challenging, time-consuming and, at least to some extent, subjective. This project will assess the role of magnetic resonance (MR) in mHE diagnosis with emphasis on multimodal imaging technique. With advanced magnetic resonance (MR) techniques, in-vivo detection of intracellular water content, estimation pH and metabolites levels with millimolar concentrations can be easily performed. This will offer to explore possible pathophysiological mechanisms of HE and to evaluate the results from previous, studies that were mainly performed on animal models or cell cultures.

By our best knowledge, multimodal MR approach as the investigators propose in this application has not been yet performed. The investigators will use advanced MR techniques which are currently not available in the clinical setting and require multicenter collaboration.

Methods The investigators will include 10-20 patients of both genders with hyperammonemia and mHE and 10-20 patients of both genders with HE. Diagnosis of HE will be made based on results of validated neuropsychiatric test. Age-matched and gender-matched control group with no gastrointestinal, neurological or psychiatric complaints and normal levels of ammonia in the blood. Patients with mHE/HE will be included from outpatient clinic of the Department of gastroenterology, University Medical Centre (UMC) Ljubljana. Healthy controls (HC) will be invited to join via internet advertisement. Contraindications for HC will include gastrointestinal (emphasis on liver disease), neurological or psychiatric complaints. Grade of mHE/HE will be classified according to West-Haven (WH) classification. Patients with different degree of liver cirrhosis, which will be scored with the Child-Pugh (CP) score, and with no contraindications for MR (e.g. presence of metal in body) will be included. Blood levels of liver enzymes and ammonia will be measured in all participants. MR scanning will include: T1- and T2-weighted MR, MRS (MEGA-PRESS and PRESS) in two voxels: striatum and cerebellum. Location will be double-checked by voxel position screenshots. Analysis, with voxel-positioning error compensation will be performed in Gannet (www.gabamrs.com). Moreover, high resolution diffusion weighted imaging (DWI), diffusion kurtosis imaging (DKI), quantitative susceptibility mapping (QSM) will be performed in brain as well. Liver QSM will be executed to assess iron load.

ELIGIBILITY:
Inclusion Criteria:

* Known liver disease/cirrhosis

Exclusion Criteria:

* Pregnancy, non compatible material with MRI

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will include 10-20 patients of both genders with signs of hepatic encephalopathy and 10-20 patients of both genders without HE. Diagnosis of HE will be made based on results of validated neuropsychiatric test. Age-matched and gender-matched control group with no gastrointestinal, neurological or psychiatric complaints and normal levels of ammonia in the blood.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Structural and Functional Changes in Brain Structures with Magnetic Resonance Imaging | 2 hours
  GABA levels and other neurotransmitters with respect to the tissue water signal and corrected for tissue composition.

CONTACTS AND LOCATIONS:
Overall Officials: Dusan Suput, M.D., Study Chair — Medical Faculty of Ljubljana; Borut Stabuc, M.D., Study Chair — Department of Gastroenterology and Hepatology, University Medical Centre Ljubljana
Locations (1):
- Department of Gastroenterology and Hepatology, University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Association for the Study of Liver Diseases; European Association for the Study of the Liver. Hepatic encephalopathy in chronic liver disease: 2014 practice guideline by the European Association for the Study of the Liver and the American Association for the Study of Liver Diseases. J Hepatol. 2014 Sep;61(3):642-59. doi: 10.1016/j.jhep.2014.05.042. Epub 2014 Jul 8. No abstract available. PMID 25015420
- [Background] Bartolic M, Vovk A, Suput D. Effects of NH4CL application and removal on astrocytes and endothelial cells. Cell Mol Biol Lett. 2016 Aug 23;21:13. doi: 10.1186/s11658-016-0011-3. eCollection 2016. PMID 28536616
- [Background] Binesh N, Huda A, Bugbee M, Gupta R, Rasgon N, Kumar A, Green M, Han S, Thomas MA. Adding another spectral dimension to 1H magnetic resonance spectroscopy of hepatic encephalopathy. J Magn Reson Imaging. 2005 Apr;21(4):398-405. doi: 10.1002/jmri.20291. PMID 15779041
- [Background] Blachier M, Leleu H, Peck-Radosavljevic M, Valla DC, Roudot-Thoraval F. The burden of liver disease in Europe: a review of available epidemiological data. J Hepatol. 2013 Mar;58(3):593-608. doi: 10.1016/j.jhep.2012.12.005. PMID 23419824
- [Background] Bustamante J, Rimola A, Ventura PJ, Navasa M, Cirera I, Reggiardo V, Rodes J. Prognostic significance of hepatic encephalopathy in patients with cirrhosis. J Hepatol. 1999 May;30(5):890-5. doi: 10.1016/s0168-8278(99)80144-5. PMID 10365817
- [Background] Chavarria L, Alonso J, Garcia-Martinez R, Simon-Talero M, Ventura-Cots M, Ramirez C, Torrens M, Vargas V, Rovira A, Cordoba J. Brain magnetic resonance spectroscopy in episodic hepatic encephalopathy. J Cereb Blood Flow Metab. 2013 Feb;33(2):272-7. doi: 10.1038/jcbfm.2012.173. Epub 2012 Nov 21. PMID 23168529
- [Background] Dale AM, Fischl B, Sereno MI. Cortical surface-based analysis. I. Segmentation and surface reconstruction. Neuroimage. 1999 Feb;9(2):179-94. doi: 10.1006/nimg.1998.0395. PMID 9931268
- [Background] Elwir S, Rahimi RS. Hepatic Encephalopathy: An Update on the Pathophysiology and Therapeutic Options. J Clin Transl Hepatol. 2017 Jun 28;5(2):142-151. doi: 10.14218/JCTH.2016.00069. Epub 2017 May 4. PMID 28660152
- [Background] Ferenci P, Lockwood A, Mullen K, Tarter R, Weissenborn K, Blei AT. Hepatic encephalopathy--definition, nomenclature, diagnosis, and quantification: final report of the working party at the 11th World Congresses of Gastroenterology, Vienna, 1998. Hepatology. 2002 Mar;35(3):716-21. doi: 10.1053/jhep.2002.31250. PMID 11870389
- [Background] Fischl B, Dale AM. Measuring the thickness of the human cerebral cortex from magnetic resonance images. Proc Natl Acad Sci U S A. 2000 Sep 26;97(20):11050-5. doi: 10.1073/pnas.200033797. PMID 10984517
- [Background] Fischl B, Salat DH, Busa E, Albert M, Dieterich M, Haselgrove C, van der Kouwe A, Killiany R, Kennedy D, Klaveness S, Montillo A, Makris N, Rosen B, Dale AM. Whole brain segmentation: automated labeling of neuroanatomical structures in the human brain. Neuron. 2002 Jan 31;33(3):341-55. doi: 10.1016/s0896-6273(02)00569-x. PMID 11832223
- [Background] Fischl B, Salat DH, van der Kouwe AJ, Makris N, Segonne F, Quinn BT, Dale AM. Sequence-independent segmentation of magnetic resonance images. Neuroimage. 2004;23 Suppl 1:S69-84. doi: 10.1016/j.neuroimage.2004.07.016. PMID 15501102
- [Background] Fischl B, Sereno MI, Dale AM. Cortical surface-based analysis. II: Inflation, flattening, and a surface-based coordinate system. Neuroimage. 1999 Feb;9(2):195-207. doi: 10.1006/nimg.1998.0396. PMID 9931269
- [Background] Fischl B, Sereno MI, Tootell RB, Dale AM. High-resolution intersubject averaging and a coordinate system for the cortical surface. Hum Brain Mapp. 1999;8(4):272-84. doi: 10.1002/(sici)1097-0193(1999)8:43.0.co;2-4. PMID 10619420
- [Background] Fischl B, van der Kouwe A, Destrieux C, Halgren E, Segonne F, Salat DH, Busa E, Seidman LJ, Goldstein J, Kennedy D, Caviness V, Makris N, Rosen B, Dale AM. Automatically parcellating the human cerebral cortex. Cereb Cortex. 2004 Jan;14(1):11-22. doi: 10.1093/cercor/bhg087. PMID 14654453
- [Background] Foerster BR, Conklin LS, Petrou M, Barker PB, Schwarz KB. Minimal hepatic encephalopathy in children: evaluation with proton MR spectroscopy. AJNR Am J Neuroradiol. 2009 Sep;30(8):1610-3. doi: 10.3174/ajnr.A1652. Epub 2009 Jun 9. PMID 19509075
- [Background] Ge PS, Runyon BA. Treatment of Patients with Cirrhosis. N Engl J Med. 2016 Aug 25;375(8):767-77. doi: 10.1056/NEJMra1504367. No abstract available. PMID 27557303
- [Background] Geissler A, Lock G, Frund R, Held P, Hollerbach S, Andus T, Scholmerich J, Feuerbach S, Holstege A. Cerebral abnormalities in patients with cirrhosis detected by proton magnetic resonance spectroscopy and magnetic resonance imaging. Hepatology. 1997 Jan;25(1):48-54. doi: 10.1053/jhep.1997.v25.pm0008985263.
- [Background] Harris AD, Saleh MG, Edden RA. Edited 1 H magnetic resonance spectroscopy in vivo: Methods and metabolites. Magn Reson Med. 2017 Apr;77(4):1377-1389. doi: 10.1002/mrm.26619. Epub 2017 Feb 2. PMID 28150876
- [Background] Hassan EA, Abd El-Rehim AS, Seifeldein GS, Shehata GA. Minimal hepatic encephalopathy in patients with liver cirrhosis: magnetic resonance spectroscopic brain findings versus neuropsychological changes. Arab J Gastroenterol. 2014 Sep-Dec;15(3-4):108-13. doi: 10.1016/j.ajg.2014.09.003. Epub 2014 Nov 11. PMID 25459346
- [Background] Haussinger D, Laubenberger J, vom Dahl S, Ernst T, Bayer S, Langer M, Gerok W, Hennig J. Proton magnetic resonance spectroscopy studies on human brain myo-inositol in hypo-osmolarity and hepatic encephalopathy. Gastroenterology. 1994 Nov;107(5):1475-80. doi: 10.1016/0016-5085(94)90552-5. PMID 7926510
- [Background] Laubenberger J, Haussinger D, Bayer S, Gufler H, Hennig J, Langer M. Proton magnetic resonance spectroscopy of the brain in symptomatic and asymptomatic patients with liver cirrhosis. Gastroenterology. 1997 May;112(5):1610-6. doi: 10.1016/s0016-5085(97)70043-x. PMID 9136840
- [Background] Lee JH, Seo DW, Lee YS, Kim ST, Mun CW, Lim TH, Min YI, Suh DJ. Proton magnetic resonance spectroscopy (1H-MRS) findings for the brain in patients with liver cirrhosis reflect the hepatic functional reserve. Am J Gastroenterol. 1999 Aug;94(8):2206-13. doi: 10.1111/j.1572-0241.1999.01228.x. PMID 10445551
- [Background] Long LL, Li XR, Huang ZK, Jiang YM, Fu SX, Zheng W. Relationship between changes in brain MRI and (1)H-MRS, severity of chronic liver damage, and recovery after liver transplantation. Exp Biol Med (Maywood). 2009 Sep;234(9):1075-85. doi: 10.3181/0903-RM-118. Epub 2009 Jun 22. PMID 19546351
- [Background] Marcellin P, Kutala BK. Liver diseases: A major, neglected global public health problem requiring urgent actions and large-scale screening. Liver Int. 2018 Feb;38 Suppl 1:2-6. doi: 10.1111/liv.13682. PMID 29427496
- [Background] Mechtcheriakov S, Schocke M, Kugener A, Graziadei IW, Mattedi M, Hinterhuber H, Vogel W, Marksteiner J. Chemical shift magnetic resonance spectroscopy of cingulate grey matter in patients with minimal hepatic encephalopathy. Neuroradiology. 2005 Jan;47(1):27-34. doi: 10.1007/s00234-004-1298-8. Epub 2005 Jan 18. PMID 15655660
- [Background] Miese F, Kircheis G, Wittsack HJ, Wenserski F, Hemker J, Modder U, Haussinger D, Cohnen M. 1H-MR spectroscopy, magnetization transfer, and diffusion-weighted imaging in alcoholic and nonalcoholic patients with cirrhosis with hepatic encephalopathy. AJNR Am J Neuroradiol. 2006 May;27(5):1019-26. PMID 16687536
- [Background] Ochoa-Sanchez R, Rose CF. Pathogenesis of Hepatic Encephalopathy in Chronic Liver Disease. J Clin Exp Hepatol. 2018 Sep;8(3):262-271. doi: 10.1016/j.jceh.2018.08.001. Epub 2018 Aug 18. PMID 30302043
- [Background] Oeltzschner G, Butz M, Baumgarten TJ, Hoogenboom N, Wittsack HJ, Schnitzler A. Low visual cortex GABA levels in hepatic encephalopathy: links to blood ammonia, critical flicker frequency, and brain osmolytes. Metab Brain Dis. 2015 Dec;30(6):1429-38. doi: 10.1007/s11011-015-9729-2. Epub 2015 Sep 11. PMID 26359122
- [Result] Albrecht J, Norenberg MD. Glutamine: a Trojan horse in ammonia neurotoxicity. Hepatology. 2006 Oct;44(4):788-94. doi: 10.1002/hep.21357. PMID 17006913